CLINICAL TRIAL: NCT00049062
Title: A Phase II And Biologic Correlative Study Investigating ARIMIDEX In Combination With IRESSA (ZD1839) In Post-Menopausal Patients With Estrogen Receptor-Positive Metastatic Breast Carcinoma Who Have Previously Failed Hormonal Therapy
Brief Title: Anastrozole and ZD 1839 in Treating Postmenopausal Women With Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000257752; CTRC-IDD-0219; CTRC-IDD-1839US; CTRC-IDD-0228
Record Dates: First submitted 2002-11-12; First posted 2003-01-27 (Estimated); Last update posted 2013-02-21 (Estimated); Status verified 2013-02

CONDITIONS: Breast Cancer
Keywords: recurrent breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Anastrozole; Gefitinib

INTERVENTIONS:
Drug: anastrozole
Drug: gefitinib

SUMMARY:
RATIONALE: Estrogen can stimulate the growth of breast cancer cells. Anastrozole may fight breast cancer by blocking the production of estrogen by the tumor cells. Biological therapies such as ZD 1839 may interfere with the growth of the tumor cells and slow the growth of advanced solid tumors. Combining anastrozole with ZD 1839 may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combining anastrozole with ZD 1839 in treating postmenopausal women who have metastatic breast cancer that has not responded to hormone therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the antitumor activity of anastrozole and ZD 1839, as measured by objective response (partial or complete) or stable disease at 6 months, in post-menopausal women with estrogen receptor-positive, hormone refractory, metastatic breast cancer.
* Determine the progression-free and overall survival of patients treated with this regimen.
* Determine the safety of this regimen in these patients.
* Determine the pharmacokinetics of this regimen in these patients.
* Correlate molecular markers with clinical benefit in patients treated with this regimen.

OUTLINE: This is an open-label, multicenter study.

Patients are stratified according to prior objective response to endocrine therapy (yes vs no).

Patients receive oral anastrozole once daily alone for 2 weeks. Patients then receive oral anastrozole and oral ZD 1839 once daily for 28 days. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Patients are followed at 1 month and then monthly thereafter.

PROJECTED ACCRUAL: A total of 36-78 patients (18-39 per stratum) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed breast cancer

  * Metastatic or locally advanced unresectable disease
* At least 1 measurable target lesion that has not been irradiated

  * New lesions in a previously irradiated field allowed as sites of measurable disease
* Progressive disease after more than 2 months of aromatase inhibitor therapy
* No known CNS disease or unevaluated CNS symptoms suggestive of brain metastases
* Hormone receptor status:

  * Estrogen receptor or progesterone receptor positive

PATIENT CHARACTERISTICS:

Age

* 18 and over

Sex

* Female

Menopausal status

* Post-menopausal by 1 of the following criteria:

  * Age 50 and over and has not menstruated during the past year or has castrate follicle-stimulating hormone (FSH) levels (greater than 40 IU/L)
  * Under age 50 and has castrate FSH levels
  * Received prior bilateral oophorectomy and has castrate FSH levels

Performance status

* ECOG 0-2

Life expectancy

* At least 12 weeks

Hematopoietic

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* ALT or AST no greater than 2.5 times ULN (5 times ULN if liver metastases present)

Renal

* Creatinine no greater than 1.5 times ULN

Cardiovascular

* No history of congestive heart failure requiring therapy
* No ventricular arrhythmia requiring therapy
* No unstable angina pectoris
* No myocardial infarction within the past 6 months

Other

* Able to swallow oral medication
* No other malignancy within the past 5 years except nonmelanoma skin cancer or carcinoma in situ of the cervix
* No known malabsorption condition or other condition that would impair absorption of study drug
* No active infection
* No other concurrent medical condition that would preclude study
* No known severe hypersensitivity to ZD 1839 or any excipients

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior chemotherapy except in adjuvant setting
* No concurrent chemotherapy for breast cancer

Endocrine therapy

* See Disease Characteristics
* More than 30 days since other prior hormonal therapy (including hormone replacement therapy and megestrol)
* Concurrent steroids for other reasons besides skin toxicity allowed
* No other concurrent hormonal therapy (including megestrol) for breast cancer

Radiotherapy

* See Disease Characteristics

Surgery

* Recovered from prior oncologic or other major surgery
* No concurrent ophthalmic surgery

Other

* More than 30 days since prior anticancer therapy
* More than 30 days since prior non-approved or investigational drugs
* No prior epidermal growth factor receptor or HER2 blockers
* No concurrent phenytoin, carbamazepine, barbiturates, rifampicin, phenobarbital, Hypericum perforatum, or systemic retinoids
* No other concurrent investigational therapy for breast cancer
* Concurrent bisphosphonates for metastatic bone disease allowed

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-09; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric K. Rowinsky, MD, Study Chair — Cancer Therapy and Research Center, Texas
Locations (1):
- Cancer Therapy and Research Center, San Antonio, Texas, United States

REFERENCES:
- [Result] Mita M, de Bono JS, Mita A, et al.: A phase II and biologic correlative study investigating anastrozole (A) in combination with geftinib (G) in post menopausal patients with estrogen receptor positive (ER) metastatic breast carcinoma (MBC) who have previously failed hormonal therapy. [Abstract] Breast Cancer Research and Treatment 94 (Suppl 1): A-1117, 2005.